CLINICAL TRIAL: NCT05325632
Title: A Phase II Study of Human Epidermal Growth Factor Receptor 2 (HER-2) Directed Dendritic Cell (DC1) Vaccine Plus Weekly Paclitaxel, Trastuzumab and Pertuzumab in Patients With HER-2 Positive Breast Cancer
Brief Title: Study of HER2 Directed Dendritic Cell (DC1) Vaccine + Weekly Paclitaxel, Trastuzumab & Pertuzumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: ImmunoRestoration (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20915
Record Dates: First submitted 2022-03-30; First posted 2022-04-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Paclitaxel; Albumin-Bound Paclitaxel; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lead In - Dose level 1 (Experimental): Six participants will be treated at dose level 1: DC vaccine given at the dose of 50 million once per week for 6 weeks
  Interventions: Biological: HER-2 pulsed DC1; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Procedure: Resection surgery
- Lead In: Dose Level 2 (Experimental): Six participants will be treated at dose level 2: DC vaccine given at the dose of 100 million once per week for 6 weeks
  Interventions: Biological: HER-2 pulsed DC1; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Procedure: Resection surgery
- Expansion -Estrogen Receptor (ER) positive (Experimental): An additional 24 participants will be enrolled at dose level 2 if determined to be safe in lead in phase to have a total of 28 evaluable participants for pathologic response assessment (including 6 pts from the lead in phase).
  Interventions: Biological: HER-2 pulsed DC1; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Procedure: Resection surgery
- Expansion -Estrogen Receptor (ER) negative (Experimental): An additional 23 participants will be enrolled at dose level 2 if determined to be safe in lead in phase to have a total of 28 evaluable participants for pathologic response assessment (including 6 pts from the lead in phase).
  Interventions: Biological: HER-2 pulsed DC1; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Procedure: Resection surgery

INTERVENTIONS:
Biological: HER-2 pulsed DC1 — Vaccine will be administered weekly for 6 weeks. Boosters will be given at months 6, 9 and 12.
Drug: Trastuzumab — 8mg/kg IV Trastuzumab will be given week 1, followed by 6 mg/kg on subsequent cycles every 3 weeks
  Other Names: Herceptin
Drug: Pertuzumab — 840 mg IV Pertuzumab will be given week 1, followed by 420 mg on subsequent cycles every 3 weeks.
  Other Names: Perjeta
Drug: Paclitaxel — 80 mg/m^2 IV paclitaxel will be given weekly weeks 7-18
  Other Names: Abraxane
Procedure: Resection surgery — After week 18, participants will undergo standard of care resection surgery.

SUMMARY:
The purpose of the study is to find out if an investigational drug called Dendritic Cell (DC1) vaccine added to standard neoadjuvant (given before main treatment) therapy can help people with HER2 (human epidermal growth factor receptor 2) positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed clinical stage I- III, HER2+ (per ASCO/CAP criteria) invasive carcinoma of the breast. Primary tumor should measure at least 1 cm by clinical exam or radiologic tests
* Candidate for neoadjuvant chemotherapy with Paclitaxel, Trastuzumab, Pertuzumab regimen followed by standard of care local therapy as determined by the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participants must have normal organ and marrow function as defined per protocol.
* Cardiac ejection fraction within institutional normal limits by either Multigated Acquisition Scan (MUGA) or Echocardiogram at baseline.
* Women of child-bearing potential and their male partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Sexually active male participants should use a barrier method or exercise abstinence during chemotherapy administration until surgery.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with inflammatory breast cancer, widespread locally advanced unresectable disease involving the chest wall/nodal basins in which a curative surgical resection cannot be performed, or those in whom de novo metastatic disease is suspected or confirmed.
* Patients may not be receiving any other investigational agents for the treatment of their breast cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study vaccine components and any of the chemotherapy drugs (paclitaxel, trastuzumab, pertuzumab).
* Participants who are unwilling or unable to undergo an apheresis for production of their vaccine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and women who are breastfeeding.
* Participants with known congenital or acquired immune deficiency (including those patients who require systemic immunosuppressant drugs for autoimmune disease or organ transplant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Lead in Phase: Immunogenicity of each dose level | at 4 weeks
  Immunogenicity: will be characterized by quantifying CD4TH1 response via ELISPot. ELISPot is an enzyme-linked immunospot assay. It is a highly sensitive immunoassay that measures the frequency of cytokine-secreting cells at the single-cell level.
Expansion Phase: Pathologic Complete Response Rate | at 12 months
  Pathologic complete response rate of participants treated in the Expansion Phase. Clinical efficacy will be defined by the pathologic complete response (pCR) rate, the percentage of patients who achieve pCR based on surgical pathology assessment. Pathologic Complete Response defined as no residual invasive disease in the breast and nodes (ypT0/is N0) at definitive surgery after completion of protocol therapy. The pathologic response to treatment will be assessed by the pathologist. The "Residual Cancer Burden" (RCB) for each patient as described in the online calculator also will be evaluated per the pathologist. (http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3)

SECONDARY OUTCOMES:
Expansion Phase: Radiologic tumor response rate after 6 weeks | at 6 weeks
  Radiologic tumor response rate measured by MRI
Expansion Phase: Radiologic tumor response rate at completion of therapy | at 12 months
  Radiologic tumor response rate measured by MRI
Expansion Phase: Immunogenicity | at 12 months
  Immunogenicity: will be characterized by quantifying CD4TH1 response via ELISPot. ELISPot is an enzyme-linked immunospot assay. It is a highly sensitive immunoassay that measures the frequency of cytokine-secreting cells at the single-cell level.
Recurrence Free Survival | up to 5 years
  Recurrence free survival defined as the length of time after treatment that patient survives without any signs or symptoms of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo (Heather) Han, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han HS, Aldrich AL, Garg SK, Weinfurtner RJ, Nguyen JV, Mo Q, Whiting J, Childress J, Soliman H, Costa R, Armaghani A, Soyano A, Kiluk J, Hoover S, Lee MC, Khakpour N, Shenoi N, Jameel Z, Koski GK, Czerniecki BJ. Alteration of the Tumor Microenvironment With Intratumoral Dendritic Cells Before Chemotherapy in ERBB2 Breast Cancer: A Nonrandomized Clinical Trial. JAMA Oncol. 2025 Feb 1;11(2):119-127. doi: 10.1001/jamaoncol.2024.5371. PMID 39636623